CLINICAL TRIAL: NCT06977256
Title: The Use of Telerehabilitation to Enhance Motor Function, Activity Performance, and Participation in Children With Developmental Coordination Disorder
Brief Title: The Use of Telerehabilitation to Improve Motor Skills and Participation in Children With Developmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10840098-772.02-4262-587
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Developmental Coordination Disorder; Telerehabilitation; Exercise; Occupational Therapy
MeSH Terms: conditions — Motor Skills Disorders; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory-Based Intervention Group (Active Comparator): For the Sensory-Based Intervention Group, participants received a 40-minute face-to-face session once a week for 8 weeks, consisting of structured exercise and sensory-based interventions. Sessions were conducted in a therapy room equipped with sensory and activity materials.
  At the end of each session, caregivers were provided with feedback, their questions were addressed, and individualized home assignments were given. The intervention program for each child was tailored to their individual needs, and the progression of activities was personalized and adjusted based on each child's performance and development throughout the study.
  Interventions: Other: Sensory-Based Exercises
- Telerehabilitation-Based Sensory Intervention Group (Experimental): For the Telerehabilitation-Based Sensory Intervention Group, participants received 40-minute in-person sensory-based sessions once a week for 8 weeks, followed by 30-minute telerehabilitation sessions once a week for an additional 8 weeks. Telerehabilitation was delivered via Zoom using a webcam-equipped computer.
  The online sessions were designed as a continuation of the face-to-face intervention and included individualized activity plans, caregiver coaching, home program recommendations, and ergonomic adjustments. Caregivers were informed in advance about required materials and setup. Each session was adapted to the child's developmental level, with activities progressively structured from simple to complex.
  Interventions: Other: Sensory-Based Exercises; Other: Telerehabilitation and Based Sensory Intervention

INTERVENTIONS:
Other: Sensory-Based Exercises — Participants in the Sensory-Based Intervention Group received weekly 40-minute face-to-face sessions for 8 weeks, involving structured exercise and sensory-based activities tailored to individual needs, with caregiver feedback and home programs provided after each session.
Other: Telerehabilitation and Based Sensory Intervention — Participants in the Telerehabilitation-Based Sensory Intervention Group received 8 weeks of in-person sessions followed by 8 weeks of weekly 30-minute telerehabilitation sessions, combining individualized sensory-based activities with caregiver coaching and home-based implementation via Zoom. Sessions were personalized, progressively structured, and conducted in a stable virtual environment to support continuity and engagement.
  Arms: Telerehabilitation-Based Sensory Intervention Group

SUMMARY:
This randomized controlled trial aimed to compare the effects of a traditional sensory-based intervention and a telerehabilitation-based sensory intervention in children aged 3-7 years diagnosed with Developmental Coordination Disorder (DCD). Participants were randomly assigned to either face-to-face or combined face-to-face and telerehabilitation groups. The outcome measures included occupational performance, sensory processing, and functional independence. The study was conducted with ethical approval, and informed consent was obtained from all legal guardians.

DETAILED DESCRIPTION:
This single-blind, parallel-group randomized controlled trial aimed to compare the effects of a traditional face-to-face sensory-based intervention and a telerehabilitation-based sensory intervention in children aged 3-7 years diagnosed with Developmental Coordination Disorder (DCD). A total of 22 participants were randomized into two groups: the Sensory-Based Intervention (SBI) group and the Telerehabilitation-Based Sensory Intervention (TBSI) group.

The SBI group received weekly 40-minute in-person sessions for 8 weeks. The TBSI group received the same 8-week in-person intervention followed by 8 weeks of weekly 30-minute telerehabilitation sessions delivered via Zoom. Both interventions included structured sensory activities tailored to each child's developmental level.

Primary and secondary outcomes were measured before and after the intervention using the Canadian Occupational Performance Measure (COPM), the Dunn Sensory Profile Parent Questionnaire, and the Functional Independence Measure for Children (WeeFIM). The study followed CONSORT guidelines and ethical approval was obtained. Written informed consent was provided by all legal guardians.

ELIGIBILITY:
Inclusion Criteria:

* Having a neurodevelopmental disorder with a confirmed diagnosis of one of the following: autism spectrum disorder, intellectual disability, developmental delay, communication disorder, or attention deficit hyperactivity disorder (ADHD)
* Absence of any condition that may interfere with cooperation during the study
* Receiving occupational therapy training for a duration between 3 months and 1 year to ensure group homogeneity in terms of prior therapy experience

Exclusion Criteria:

* Presence of any visual or hearing impairment that could affect study outcomes
* Having any systemic disease
* Having a physical disability that may interfere with movement or motor function

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | From enrollment to the end of treatment at 8 weeks
  The Canadian Occupational Performance Measure (COPM) is a standardized assessment tool frequently used by occupational therapists to identify problems in occupational performance areas and to measure individuals' perceived performance and satisfaction levels. The COPM is administered through a semi-structured interview and takes approximately 20-30 minutes to complete. It involves individuals rating their performance and satisfaction in the areas of self-care, productivity, and leisure activities. The COPM has been adapted and validated across various age groups and diagnostic populations and is commonly used in pediatric settings as well.
Dunn Sensory Profile | From enrollment to the end of treatment at 8 weeks
  In this study, the Parent Questionnaire version of the Sensory Profile was administered to assess the sensory processing patterns of participating children. Developed by Winnie Dunn in 1999, the Sensory Profile is designed for children aged 3 to 10 and consists of 125 items evaluating various aspects of sensory development. The tool identifies four sensory response patterns: sensitivity, registration, avoidance, and seeking. Scoring is categorized into three main domains: sensory processing, modulation, and behavioral/emotional responses. The questionnaire includes subscales such as auditory, visual, vestibular, tactile, multisensory, and oral sensory processing, as well as items addressing endurance, posture, activity level, emotional modulation, and social-emotional responses.
Functional Independence Measure for Children (WeeFIM) | From enrollment to the end of treatment at 8 weeks
  The Functional Independence Measure for Children (WeeFIM) was developed to address the sensitivity and comprehensiveness limitations of the Barthel Index in assessing functional independence. It evaluates both motor and cognitive components of a child's functional abilities and is based on the International Classification of Functioning, Disability and Health (ICF). The WeeFIM consists of 18 items, divided into two domains: 13 items in the motor domain and 5 items in the cognitive domain. It is commonly used to assess the level of assistance required by children in daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Mazlum Uruc, MSc, Principal Investigator — Medipol University
Locations (1):
- Günışığı Counseling Center and Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

REFERENCES:
- [Derived] Uruc M, Menek B. The effect of telerehabilitation on activity performance and participation in daily life in children with developmental coordination disorder: A randomized controlled trial. PLoS One. 2025 Aug 21;20(8):e0330846. doi: 10.1371/journal.pone.0330846. eCollection 2025. PMID 40839575